CLINICAL TRIAL: NCT01374269
Title: Improvement in Pain, Function and Quality of Life With a Protocolized Exercise Program Compared With Non-steroidal Anti-inflammatory Analgesics in Patients With Subacute Low Back Pain in Medellín, Colombia, 2009-2010
Brief Title: Improvement in Pain,Function and HRQoL ( Health Related Quality of Life) in Subacute Low Back Pain: A Controlled Clinical Trial of Exercise vs NSAIDs (Nonsteroidal Antiinflammatory)
Acronym: DLSEA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grupo Rehabilitacion en Salud (Network)
Collaborators: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Fabio Alonso Salinas Duran, Associate Professor, Grupo Rehabilitacion en Salud
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DLSejervsaine; DLSEjercicioyAINES (Registry Identifier: GrupoRS)
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-03

CONDITIONS: Back Pain Lower Back
Keywords: NSAIDS (Nonsteroidal anti-inflammatory drugs); Exercise; Physiotherapy; Subacute Low Back Pain; Pain; Visual Analogue Scale; oswesrty; Roland Morris; SF-36; Quality of life
MeSH Terms: conditions — Low Back Pain; Motor Activity; Pain | interventions — Resistance Training; Exercise Therapy; Physical Therapy Modalities; Anti-Inflammatory Agents, Non-Steroidal; Naproxen; Celecoxib; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Excercise (Experimental): One group will be assigned to protocolized back pain exercise, three times a week for 4 weeks. This program is carried out by physiotherapists from participating institutions who wish to participate in research and who will be given a training which will standardize the intervention programs Exercise program includes: physical agents, massage of myofascial points, stretching and strengthening exercises, cycloergometer or band aerobic exercises. Treatment, type of exercises, exercise tolerance and adverse reactions will be registered
  Interventions: Other: Exercise program
- NSAID (Active Comparator): Naproxen 500 mg per day by 10 days or Celecoxib 200 mg per day by 10 days and Acetaminophen 1,5 a 2 g as rescue
  Interventions: Drug: NSAID (Nonsteroidal anti-inflammatory drugs)

INTERVENTIONS:
Other: Exercise program — Standardize the intervention programs Exercise program includes: physical agents, massage of myofascial points, stretching and strengthening exercises, cycloergometer or band aerobic exercises. 12 sessions, 3 per week.
  Other Names: Therapeutic exercise; Physiotherapy
  Arms: Excercise
Drug: NSAID (Nonsteroidal anti-inflammatory drugs) — The second group was treated for 10 days with NSAIDs (naproxen 500 mg/d or celecoxib 200 mg/d) according to the indications and contraindications. The patients kept a journal stating whether they had taken the drug and any adverse reactions. If the pain intensity of any participant increased, acetaminophen (1.5 - 2.0 g/d) was proposed as a rescue procedure.
  Other Names: Naproxen; Celecoxib; Acetaminophen
  Arms: NSAID

SUMMARY:
Our clinical trial has the purpose to evaluate the effectiveness in reducing pain and improving function and quality of life during a 6-months follow-up of a therapeutic exercise program compared to pharmacological treatment with NSAIDs in patients with subacute low back pain attending the physiatrist consultation of several ambulatory health centers in Medellín during the years 2009-2010.

DETAILED DESCRIPTION:
General Purpose To evaluate the effectiveness in reducing pain and improving function and quality of life during a 6-months follow-up of a therapeutic exercise program compared to pharmacological treatment with NSAIDs in patients with subacute low back pain attending the physiatrist consultation of several ambulatory health centers in Medellín during the years 2009-2010.

Specific Objectives

1. To evaluate the efficacy of a protocolized exercise program in reducing low back pain.
2. To evaluate the efficacy of a protocolized exercise program in improving the function.
3. To compare the effects of both interventions on quality of life and work absenteeism in the two groups of patients.
4. To compare the safety of both interventions.
5. To estimate adherence and causes of non-adherence of patients to different treatments proposed.
6. To compare in both groups the number of relapses, general and specialized medical consultations, screening studies, images and other treatments associated with low back pain.

   Null Hypothesis Management of subacute low back pain patients with a protocolized exercise program is not more effective than treatment with NSAIDs to reduce pain at least in 25 mm, measured with a Visual Analog Scale 0-100 mm.

   Alternative hypothesis Management of subacute low back pain patients with a protocolized exercise program is not more effective than treatment with NSAIDs to reduce pain at least in 25 mm, measured with a Visual Analog Scale 0-100 mm.

   Methodology:

   Type of study: randomized controlled clinical trial, single-blinded with independent evaluators.

   Reference population: Patients consulting physiatrists in different physical medicine and rehabilitation departments in Medellin, Colombia.

   Study population: patients with subacute low back pain -evolution time more than 6 weeks and less than 3 months-, with or without radiculopathy, and that fulfill inclusion criteria. In addition patients must sign an informed consent to participate in research.

   Inclusion criteria:
   * Patients aged between 18 and 60 years with subacute low back pain.
   * Evolution time more than 6 weeks and less than 3 months.
   * That were included in the social security system and live in the metropolitan area.

   Exclusion criteria:
   * Antecedents of spinal, pelvis or abdominal trauma.
   * Cancer.
   * Diabetes mellitus.
   * Steroid use.
   * Women over 60 years.
   * Cauda equine syndrome.
   * Men with osteoporosis or compression fractures.
   * Suspicion of infection
   * Insidious onset
   * Constitutional symptoms
   * Intravenous drugs abuse
   * HIV
   * Immunosuppression
   * Previous surgery
   * Rheumatic diseases
   * Urinary tract infections
   * Neurological symptoms in lower limbs
   * Mental illness (schizophrenia, bipolar or somatomorphic disorder, major depression)
   * Deformities in the spine (scoliosis greater than 15º)
   * History of peptic acid disease
   * Renal failure
   * Intake of anticoagulants or antiplatelet drugs
   * Allergy to NSAIDs.

   Primary outcome Pain relief more than 25 mm on the Visual Analogue Scale, ranging from 0 to 100, assessed 4 weeks after intervention.

   Secondary outcomes:

   Improvement in function assessed by the Oswestry Disability Index and Roland-Morris questionnaire comparing baseline to first, three and six months follow-up.

   Improvement in quality of life assessed by SF-36 (The Short Form Health Survey) questionnaire at baseline and at first, third and sixth months.

   Work absenteeism decrease. Decrease in the number of relapses, general and specialized medical consultations, screening studies, images and other treatments associated with low back pain at 6 months.

   Safety of both treatments evaluated in the exercise group by tolerance to training and presence or not of side effects, and in the NSAIDs group by the presence or absence of adverse reactions.

   Sample:

   Sampling type: simple random. Sample size calculation was based on software "Sample size Javeriana University" Type I error: 0.05 Type II Error: 0.2 Assessments number prior to randomization: 1 Assessments number after randomization: 3 Correlation between evaluations: 0.8 Clinically important difference: 0.33 Number of patients per group: 33 Experimental group control group ratio : 1 to 1 10% of loss: 7 Total: 73

   Randomization Randomization was done by means of permuted blocks of size 2, 4 and 6, generated by computer (Ralloc program, co Stata 8.2, College Station, TX, USA). Allocation will be confidential and will not be opened until the investigation is completed, this will be monitored by the Committee of Data Security.

   Enrollment Patients with subacute low back pain consulting Physical Medicine and Rehabilitation Departments of hospitals in Medellín, Colombia. There will be an initial assessment, and if patient is considered eligible will be invited to participate and asked to sign an informed consent (Appendix 1). Treatment assignment will be given in an opaque envelope.

   Masking Medical researchers who evaluate the patients, research assistants who perform the application of different measure instruments and statistical will be blinded to treatment allocation.

   Initial assessment Clinical evaluation will be performed by one of the research physiatrists. Evaluation will include: epidemiological and clinical, Visual Analog Scale (VAS), Oswestry scale, Rolland Morris Scale, and SF-36 quality of life scale.

   Intervention One group will be assigned to protocolized back pain exercise, three times a week for 4 weeks. This program is carried out by physiotherapists from participating institutions who wish to participate in research and who will be given a training which will standardize the intervention programs Exercise program includes: physical agents, massage of myofascial points, stretching and strengthening exercises, cycloergometer or band aerobic exercises. Treatment, type of exercises, exercise tolerance and adverse reactions will be registered. The second group will receive NSAID for 10 days, there will be two different options (naproxen or celecoxib) according to indications and contraindications. In case of increase in pain intensity in either of the two groups, acetaminophen in doses of 1.5 to 2.0 g / day will be used as a rescue.

   Adherence to different treatments. To ensure adherence to different treatments each patient will receive a phone call weekly to inquire about assistance, difficulties, tolerance, use of medications, and adverse effects. Patients will be given a questionnaire to verify drugs intake, dosage, time and side effects. They should also register any other drug ingestion.

   Telephone calls will be made every 15 days to ask about the health status and ensuring assistance to new assessments.

   Assessment will be scheduled at 1, 3, and 6 months Clinical evaluation will be performed by one of the researcher physiatrists or a postgraduate student.

   Committee of safety and quality of data. This committee will consist of two researchers and one professional information management responsible for the database. This will be done in Access and SPSS 15 (Statistical Product and Service Solutions) before starting information recollection.

   Analysis Plan Categorical univariate variables will be analyzed by frequency distributions and quantitative variables by measures of central tendency (mean, standard deviation, median or range). Both groups will be compared after randomization and before intervention for all variables.

   Initially, it will be established for each group if the quantitative variables are of normal distribution, by using the Kolmogorov-Smirnov test.

   Pain (primary outcome) will be evaluated in each patient at 1, 3 and 6 months and will be compared with initial pain (mean and confidence intervals) by using Student t test or Mann Whitney for each time period. The same procedure would be for the other outcomes measured quantitatively.

   An analysis of variance with repeated measures for the variability between groups and intragroup will be made.

   Comparison of categorical variables at each assessment will be done using the Chi2 test.

   The level of statistical significance to be used in all cases is 0.05. An analysis by intention to treat and per protocol will be made.

   Ethics This research and informed consent is according to "Scientific, technical and administrative standards for health research" of the Ministry of Health and the Decree 309 of 2000 of the Ministry of Environment. This is considered a minimal risk research, because therapeutic interventions are widely used to treat patients with these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 60 years old
* Subacute low back pain -evolution time more than 4 weeks and less than 3 months.
* That have social security system
* Live in the metropolitan area

Exclusion Criteria:

* Antecedents of spinal, pelvis or abdominal trauma
* Cancer
* Diabetes mellitus
* Steroids use
* Men and Women over 60 years
* Cauda equine syndrome
* Women and men with osteoporosis or compression fractures
* Suspicion of infection.
* Insidious onset, constitutional symptoms
* Intravenous drugs abuse
* HIV
* Immunosuppression or previous surgery
* Rheumatic diseases
* Urinary tract infections
* Neurological symptoms in lower limbs
* Mental illness (schizophrenia, bipolar or somatomorphic disorder, major depression)
* Deformities in the spine (scoliosis greater than 15º)
* History of peptic acid disease
* Renal failure
* Intake of anticoagulants or antiplatelet drugs
* Allergy to NSAIDs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luz H Lugo, Professor, Study Director — Universidad de Antioquia
Locations (2):
- Colombia (2):
  - Clínica de Las Américas, Medellín, Antioquia
  - Ips Universitaria, Medellín, Antioquia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients (18 and 60 years) with SLBP (subacute low back pain) (lasting 4-12 weeks) with or without radiculopathy who were assigned to the social security system and living in the metropolitan area were included.
Pre-assignment Details: A specific cause for the pain (infection, tumor, ankylosing spondylitis, inflammatory conditions or cauda equine syndrome), the presence of red flags, scoliosis >15 °, depression or mental illness, history of gastrointestinal bleeding, renal failure, intake of anticoagulants or antiplatelet drugs and NSAID allergy were excluded.
Groups:
- Excercise: One group will be assigned to protocolized back pain exercise, three times a week for 4 weeks. This program is carried out by physiotherapists from participating institutions who wish to participate in research and who will be given a training which will standardize the intervention programs Exercise program includes: physical agents, massage of myofascial points, stretching and strengthening exercises, cycloergometer or band aerobic exercises. Treatment, type of exercises, exercise tolerance and adverse reactions will be registered
  Exercise program : Standardize the intervention programs Exercise program includes: physical agents, massage of myofascial points, stretching and strengthening exercises, cycloergometer or band aerobic exercises. 12 sessions, 3 per week.
- NSAID: Naproxen 500 mg per day by 10 days or Celecoxib 200 mg per day by 10 days and acetaminophen 1,5 a 2 g as rescue
  NSAID : The second group was treated for 10 days with NSAIDs (naproxen 500 mg/d or celecoxib 200 mg/d) according to the indications and contraindications. The patients kept a journal stating whether they had taken the drug and any adverse reactions. If the pain intensity of any participant increased, acetaminophen (1.5 - 2.0 g/d) was proposed as a rescue procedure.
Period: Overall Study
Arm/Group | Excercise | NSAID
Started | 46 | 44
Completed | 40 | 39
Not Completed | 6 | 5
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — closed research | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Excercise | NSAID | Total
Number analyzed (Participants) | 46 | 44 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (12.3) | 40.3 (13.2) | 39.4 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 70
  Male | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  Colombia | 46 | 44 | 90

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale of Pain
Description: In the Visual Analogue Sacale the best result is 0 and the worst is 100, The primary outcome was pain the mesurement of the Visual Analog Scale (VAS) (0 [no pain] to 100 [maximum pain]) at the beginning.
Time Frame: At the beginning
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 47.3 (19.8) | 45.2 (22.6)

2. Secondary Outcome: Oswestry Disability Index
Description: Function was assessed using the Oswestry Disability Index questionnaire Version 2.1a, which ranges from 0 to 100 (greater disability), being worst 100. The Oswestry Disability Index is currently considered by many as the gold standard for measuring degree of disability and estimating quality of life in a person with low back pain. 0% to 20%: Minimal disability, 21%-40%: Moderate Disability, 41%-60%: Severe Disability, 61%-80%: Crippling back pain, 81%-100%: These patients are either bed-bound or have an exaggeration of their symptoms.
Time Frame: At the beginning
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 28.9 (13.1) | 29.4 (15.1)

3. Secondary Outcome: Oswestry Disability Index
Description: as for outcome 2
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 21.9 (12.6) | 26.6 (18.5)

4. Secondary Outcome: Oswestry Disability Index
Description: as for outcome 2
Time Frame: 12 weeks
Population: We lost 4 patients in arm exercise because we ran out of time limit for the investigation and could not evaluate them. And we lost 4 in arm NSAIDs, 3 who did not answer our calls and 1 for close investigation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
units on a scale | 16.6 (13.2) | 19.4 (13.7)

5. Secondary Outcome: Oswestry Disability Index
Description: as for outcome 2
Time Frame: 24 weeks
Population: We lost 2 patients in arm exercise 1 because we ran out of time limit for the investigation and could not evaluate them and 1 who did not answer our calls . In the NSAIDs arm we recover 3 patients who did not answer the call for three months evaluation, and lost 4 for deadline of the investigation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
units on a scale | 13.8 (12.2) | 17.2 (14.0)

6. Secondary Outcome: Roland-Morris Questionnaire
Description: Improvement in function assessed by the Roland-Morris questionnaire, a widely used health status measure for low back pain. The RMDQ can be used in research or clinical practice. Scoring the RMDQ. The RMDQ is scored by adding up the number of items checked by the patient. The score can therefore vary from 0 to 24. It is not recommended to give patients a 'Yes' / 'No' option. If patients indicate in any way that an item is not applicable to them, the item is scored 'No', i.e. the denominator remains 24. Being worst 24.
Time Frame: At the beginning
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 6.9 (4.4) | 7.7 (5.2)

7. Secondary Outcome: Roland-Morris Questionnaire
Description: as for outcome 6
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 4.2 (3.2) | 4.6 (4.0)

8. Secondary Outcome: Roland-Morris Questionnaire
Description: as for outcome 6
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
units on a scale | 2.6 (2.5) | 3.2 (2.4)

9. Secondary Outcome: Roland-Morris Questionnaire
Description: as for outcome 6
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
units on a scale | 2.3 (3.0) | 2.5 (2.6)

10. Secondary Outcome: Quality of Life, Change in Health
Description: Improvement in Quality of life was assessed with the SF-36 questionnaire, which ranges from 0 to 100 being 100 the best quality of life. The Short Form (36) Health Survey is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e. a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. This outcome shows the subdomain data: change in health.
Time Frame: At the beginning
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 52.6 (13.5) | 54.5 (16.9)

11. Primary Outcome: Visual Analogue Scale of Pain
Description: In the VAS the best result is 0 and the worst is 100. The primary outcome was pain improvement of ≥25 mm on the Visual Analog Scale (VAS) (0 [no pain] to 100 [maximum pain]) at 4 weeks.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 28.8 (20.5) | 34.9 (25.0)

12. Primary Outcome: Visual Analogue Scale of Pain
Description: In the VAS the best result is 0 and the worst is 100. The primary outcome was pain improvement of ≥25 mm on the Visual Analog Scale (VAS) (0 [no pain] to 100 [maximum pain]) at 12 weeks.
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
units on a scale | 21.0 (24.4) | 20.6 (17.2)

13. Primary Outcome: Visual Analogue Scale of Pain
Description: The best result is 0 and the worst is 100, Pain relief more than 25 mm on the Visual Analogue Scale, assessed 24 weeks after intervention.
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
units on a scale | 17.8 (21.8) | 17.5 (18.1)

14. Secondary Outcome: Quality of Life, Change in Health
Description: as for outcome 10
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 60.4 (18.1) | 61.3 (21.7)

15. Secondary Outcome: Quality of Life, Change in Health
Description: as for outcome 10
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
units on a scale | 73.3 (21.0) | 67.0 (20.5)

16. Secondary Outcome: Quality of Life, Change in Health
Description: as for outcome 10
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
units on a scale | 78.0 (18.0) | 70.7 (18.2)

17. Secondary Outcome: Quality of Life, Bodily Pain
Description: Improvement in Quality of life was assessed with the SF-36 questionnaire, which ranges from 0 to 100 being 100 the best quality of life. The Short Form (36) Health Survey is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e. a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. This outcome shows the subdomain data: bodily pain.
Time Frame: At the beginning
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 39.5 (13.4) | 39.2 (13.3)

18. Secondary Outcome: Quality of Life, Bodily Pain
Description: as for outcome 17
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 57.8 (18.7) | 54.0 (19.5)

19. Secondary Outcome: Quality of Life, Bodily Pain
Description: as for outcome 17
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
units on a scale | 67.6 (21.7) | 58.7 (16.1)

20. Secondary Outcome: Quality of Life, Bodily Pain
Description: as for outcome 17
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
units on a scale | 74.1 (22.4) | 68 (20.6)

21. Secondary Outcome: Quality of Life, Emotional Performance.
Description: Improvement in Quality of life was assessed with the SF-36 questionnaire, which ranges from 0 to 100 being 100 the best quality of life. The Short Form (36) Health Survey is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e. a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. This outcome shows the subdomain data: Emotional Performance.
Time Frame: At the beginning
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 67.2 (36.6) | 63.4 (38.4)

22. Secondary Outcome: Quality of Life, Emotional Performance.
Description: as for outcome 21
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 82.5 (32.8) | 84.7 (29.2)

23. Secondary Outcome: Quality of Life, Emotional Performance.
Description: as for outcome 21
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
units on a scale | 91.2 (24.5) | 82.4 (33.8)

24. Secondary Outcome: Quality of Life, Emotional Performance.
Description: as for outcome 21
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
units on a scale | 94.1 (21.2) | 93.9 (20.1)

25. Secondary Outcome: Quality of Life, Physical Performance.
Description: Improvement in Quality of life was assessed with the SF-36 questionnaire, which ranges from 0 to 100 being 100 the best quality of life. The Short Form (36) Health Survey is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e. a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. This outcome shows the subdomain data: Physical Performance
Time Frame: At the beginning
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 30.5 (34.0) | 36.0 (40.9)

26. Secondary Outcome: Quality of Life, Physical Performance.
Description: as for outcome 25
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 58.1 (39.4) | 55.1 (42.9)

27. Secondary Outcome: Quality of Life, Physical Performance.
Description: as for outcome 25
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
units on a scale | 77.3 (33) | 72.5 (40.7)

28. Secondary Outcome: Quality of Life, Physical Performance.
Description: as for outcome 25
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
units on a scale | 84.3 (33.3) | 85.2 (30.7)

29. Secondary Outcome: Quality of Life, Physical Function.
Description: Improvement in Quality of life was assessed with the SF-36 questionnaire, which ranges from 0 to 100 being 100 the best quality of life. The Short Form (36) Health Survey is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e. a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. This outcome shows the subdomain data: Physical Function.
Time Frame: At the beginning
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 64.6 (21.6) | 66.5 (17.8)

30. Secondary Outcome: Quality of Life, Physical Function.
Description: as for outcome 29
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 75.8 (17.5) | 70.3 (23.3)

31. Secondary Outcome: Quality of Life, Physical Function.
Description: as for outcome 29
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
units on a scale | 81.6 (16) | 77.2 (82.6)

32. Secondary Outcome: Quality of Life, Physical Function.
Description: as for outcome 29
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
units on a scale | 84.1 (16.9) | 82.6 (16.0)

33. Secondary Outcome: Quality of Life, Social Function.
Description: Improvement in Quality of life was assessed with the SF-36 questionnaire, which ranges from 0 to 100 being 100 the best quality of life. The Short Form (36) Health Survey is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e. a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. This outcome shows the subdomain data: Social Function.
Time Frame: At the beginning
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 71.3 (23.5) | 65.9 (24.2)

34. Secondary Outcome: Quality of Life, Social Function.
Description: as for outcome 33
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 80.7 (19.9) | 74.8 (24.4)

35. Secondary Outcome: Quality of Life, Social Function.
Description: as for outcome 33
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
units on a scale | 87.3 (17.2) | 80.4 (18.3)

36. Secondary Outcome: Quality of Life, Social Function.
Description: as for outcome 33
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
units on a scale | 88.6 (17.4) | 86 (15.1)

37. Secondary Outcome: Quality of Life, General Health Perceptions.
Description: Improvement in Quality of life was assessed with the SF-36 questionnaire, which ranges from 0 to 100 being 100 the best quality of life. The Short Form (36) Health Survey is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e. a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. This outcome shows the subdomain data: General Health Perceptions.
Time Frame: At the beginning
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 64.3 (19.1) | 64.7 (18.3)

38. Secondary Outcome: Quality of Life, General Health Perceptions.
Description: as for outcome 37
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 66.3 (18.5) | 67.1 (20.01)

39. Secondary Outcome: Quality of Life, General Health Perceptions.
Description: as for outcome 37
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
units on a scale | 72.0 (19.9) | 69.2 (16.9)

40. Secondary Outcome: Quality of Life, General Health Perceptions.
Description: as for outcome 37
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
units on a scale | 73.4 (17.6) | 69.3 (15.8)

41. Secondary Outcome: Quality of Life, Mental Health.
Description: Improvement in Quality of life was assessed with the SF-36 questionnaire, which ranges from 0 to 100 being 100 the best quality of life. The Short Form (36) Health Survey is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e. a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. This outcome shows the subdomain data: Mental Health.
Time Frame: At the beginning
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 66.4 (20.6) | 67.0 (19.8)

42. Secondary Outcome: Quality of Life, Mental Health.
Description: as for outcome 41
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 71.4 (18.9) | 74.6 (20.0)

43. Secondary Outcome: Quality of Life, Mental Health.
Description: as for outcome 41
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
units on a scale | 76.4 (16.4) | 75.6 (16.5)

44. Secondary Outcome: Quality of Life, Mental Health.
Description: as for outcome 41
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
units on a scale | 78.5 (16.1) | 76.9 (16.3)

45. Secondary Outcome: Quality of Life, Vitality.
Description: Improvement in Quality of life was assessed with the SF-36 questionnaire, which ranges from 0 to 100 being 100 the best quality of life. The Short Form (36) Health Survey is a patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e. a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. This outcome shows the subdomain data: Vitality.
Time Frame: At the beginning
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 55.5 (17.9) | 55.3 (17.6)

46. Secondary Outcome: Quality of Life, Vitality.
Description: as for outcome 45
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 61.3 (18.5) | 64.0 (20.2)

47. Secondary Outcome: Quality of Life, Vitality.
Description: as for outcome 45
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
units on a scale | 67.5 (17.7) | 66.6 (15.6)

48. Secondary Outcome: Quality of Life, Vitality.
Description: as for outcome 45
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
units on a scale | 70.3 (17.0) | 62.8 (14.5)

49. Secondary Outcome: PHQ-9 Patient Health Questionnaire (PHQ-9) Depression
Description: Depression was measured with the Patient Health Questionnaire (PHQ-9), which ranged from 0 (no depression) to 27 (severe depression).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 3.9 (4.0) | 3.4 (3.3)

50. Secondary Outcome: PHQ-9 Patient Health Questionnaire (PHQ-9) Depression
Description: as for outcome 49
Time Frame: At the beginning
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
units on a scale | 5.7 (4.3) | 5.1 (3.0)

51. Secondary Outcome: PHQ-9 Patient Health Questionnaire (PHQ-9) Depression
Description: as for outcome 49
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
units on a scale | 3.0 (3.1) | 3.2 (2.7)

52. Secondary Outcome: PHQ-9 Patient Health Questionnaire (PHQ-9) Depression
Description: as for outcome 49
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
units on a scale | 2.3 (2.5) | 3.1 (3.0)

53. Secondary Outcome: Relapses of Lumbar Pain
Description: The percentage of patients with relapsed of low back pain was measured.
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
percentage of participants | 7.1 | 25

54. Secondary Outcome: Relapses of Lumbar Pain
Description: The percentage of patients with relapsed of low back pain was measured.
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
percentage of participants | 5.0 | 20.5

55. Secondary Outcome: Treatments Associated With Low Back Pain at 6 Months
Description: we are showing in this result, the number of patients who had to receive any additional treatment in either group. The measure is the number of participants who received additional treatment throughout the duration of the study.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
participants | 3 | 14

56. Secondary Outcome: Missing Workdays
Description: This result shows the average of the number of missed work days.
Time Frame: 6 weeks before starting
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
Days | 1.0 (2.9) | 1.7 (6.2)

57. Secondary Outcome: Missing Workdays
Description: This result shows the average of the number of missed work days.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
Days | 0.0 (0.0) | 0.3 (1.6)

58. Secondary Outcome: Missing Workdays
Description: This result shows the average of the number of missed work days.
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
Days | 0.0 (0.4) | 0.1 (0.6)

59. Secondary Outcome: Missing Workdays
Description: This result shows the average of the number of missed work days.
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
Days | 0.2 (0.7) | 0.2 (0.9)

60. Secondary Outcome: Medical Consultations.
Description: This result shows, the total number of participants received additional medical consultations.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 46 | 44
participants | 4 | 6

61. Secondary Outcome: Medical Consultations.
Description: This result shows, the total number of participants received additional medical consultations.
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 42 | 40
participants | 1 | 6

62. Secondary Outcome: Medical Consultations.
Description: This result shows, the total number of participants received additional medical consultations.
Time Frame: 24 weeks
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Excercise | NSAID
Number analyzed (Participants) | 40 | 39
participants | 4 | 4

ADVERSE EVENTS:
Time Frame: Adverse effects were recorded that occurred during the 6-month study
Arm/Group | Excercise | NSAID
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/44
Other Adverse Events (participants affected / at risk) | 0/46 | 14/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Excercise (N=46) | NSAID (N=44)
Epigastric pain (Gastrointestinal disorders) | 0 (0) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 5 (5)
Rash (Immune system disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The study population was associated with the university's health service. Female subjects predominated. The 6-month follow-up prevents conclusions about the improvement duration. No subgroup classification was performed. No control group was planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No